CLINICAL TRIAL: NCT00621413
Title: Dosimetric and Morbidity Outcomes of Cs-131 Brachytherapy in Combination With External Beam Radiation Therapy in Subjects With Intermediate to High Risk Adenocarcinoma of the Prostate: An Observational Study
Brief Title: Observation of Outcomes and Side Effects of Cesium-131 in Combination With External Beam Radiation for the Treatment of Intermediate to High Risk Prostate Cancer
Status: Withdrawn | Type: Observational
Why Stopped: Study never moved forward due to no accrual
Sponsor: IsoRay Medical, Inc. (Industry)
Collaborators: Swedish Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: isoray_cs131_pc01
Record Dates: First submitted 2008-02-12; First posted 2008-02-22 (Estimated); Last update posted 2021-04-19 (Actual); Status verified 2021-04

CONDITIONS: Prostate Cancer
Keywords: prostate; cancer; intermediate risk; high risk; brachytherapy; Cesium-131; seed brachytherapy; intermediate and high risk cancer of the prostate
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to observe PSA response and incidence of side effects in patients diagnosed with intermediate to high risk prostate cancer and treated with Cesium-131 in combination of external beam therapy.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed adenocarcinoma of the prostate
* Clinical stage T1c - T2c (AJCC 6th Edition), NX/N0, M0
* Karnofsky Performance Score of 90 to 100
* Greater than or equal to 18 years of age
* Prostate volumes by TRUS ≤ 60 cc
* I-PSS score < 15 (alpha blockers allowed)
* Signed study-specific informed consent form prior to study entry

Intermediate Risk prostate cancer as determined by the following:

* Gleason sum of 7; PSA less than 10.1 ng/ml; Stage T2a or less
* Gleason sum 6 or less; PSA >10.0 and < 20.1ng/ml; Stage T2a or less
* Gleason sum 6 or less; PSA < 10.1; Stage T2b

High risk prostate cancer as determined by the following:

* Any Gleason Sum; PSA greater than 20 ng/ml; Stage T2c or less
* Gleason Sum > 7; Any PSA; Stage T2c or less
* Any Gleason Sum; Any PSA; Stage T2c
* Any two or three intermediate risk factor

Exclusion Criteria:

* Lymph node involvement (N1)
* Evidence of distant metastases (M1)
* Any hormonal blockade or therapy that:

  * Has persisted for more than 6 months by time of protocol screening; OR
  * Is ongoing within 3 months of study enrollment
* Radical surgery for carcinoma of the prostate
* Prior pelvic radiation
* Previous or concurrent cancers other than basal, in situ, or squamous cell skin cancers unless disease-free for ≥ 5 years
* Major medical or psychiatric illness, which in the investigator's opinion, would prevent completion of treatment and would interfere with follow-up
* Hip prosthesis
* Inability or refusal to provide informed consent

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: diagnosed patients with intermediate to high risk cancer of the prostate. Patient will be in a Radiation Oncology setting.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2007-02 (Estimated); Primary Completion 2007-02 (Actual); Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
The analysis of dosimetric data resultant from Cs-131 permanent prostate brachytherapy in combination with external beam radiation therapy in the setting of intermediate to high risk cancer of the prostate. | 5 years
  Data collected for analysis will be total therapeutic dose delivered to the prostate by the Cs-131 brachytherapy implant treatment in units of Gy.

SECONDARY OUTCOMES:
The analysis of treatment related morbidities following Cs-131 prostate brachytherapy in combination with external beam therapy for intermediate to high risk cancer of the prostate. | 5 years
  Data collected for analysis will be the EPIC prostate cancer quality of life questionnaire.
The analysis of PSA control rates following Cs-131 prostate brachytherapy in combination with external beam therapy for intermediate to high risk cancer of the prostate. | 5 years
  Data collected for analysis will be PSA measurements.

CONTACTS AND LOCATIONS:
Overall Officials: John Sylvester, MD, Principal Investigator — Seattle Prostate Institute / Swedish Hospital; Steve Kurtzman, MD, Principal Investigator — Mills Peninsula Hospital
Locations (9):
- United States (9):
  - Arizona Oncology Services Foundation, Phoenix, Arizona
  - Eisenhower Medical Center, Rancho Mirage, California
  - Dorthory Schneider Cancer Center, San Mateo, California
  - Levine Cancer Center, Worcester, Massachusetts
  - St. Mary's Regional Medical Center, Reno, Nevada
  - Northshore Medical Accelerator, Smithtown, New York
  - Sentara Cancer Institute, Hampton, Virginia
  - Virginia Mason Medical Center, Seattle, Washington
  - Seattle Prostate Institute / Swedish Hospital, Seattle, Washington